CLINICAL TRIAL: NCT02789098
Title: Assessment of Coronary Endothelial Function and Myocardial Fibrosis in Positron Emission Tomography With the Waning of Acute Coronary Syndrome With Elevated ST Segment : Relationship With Left Ventricular Remodeling
Brief Title: Relationship Between Left Ventricular Remodeling, Coronary Endothelial Function and Myocardial Fibrosis Using Positron Emission Tomography in Patients With ST-elevation Myocardial Infarction
Acronym: REMOD-TEP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical issues.
Sponsor: University Hospital, Caen (Other)
Collaborators: Société Française de Cardiologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-A01650-49
Record Dates: First submitted 2016-04-21; First posted 2016-06-02 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST Elevation Myocardial Infarction; Ventricular remodeling; Biomarkers; Coronary endothelial function; Positron Emission Tomography
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ventricular Remodeling | interventions — Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STEMI (Other): All patients included in this study (1 arm)
  Interventions: Other: (15)-O water positron emission tomography and Biomarkers

INTERVENTIONS:
Other: (15)-O water positron emission tomography and Biomarkers — Coronary endothelial function is assessed using (15)-O water positron emission tomography and cold pressor test . The response to the test is defined by the percentage increase myocardial blood flow . Assessment of fibrosis, inflammation an endothelial function is performed using biomarkers.

SUMMARY:
Left ventricular remodeling is a common complication in patients with ST-elevation myocardial infarction (STEMI ) and may lead to heart failure. Hemodynamic, metabolic and inflammatory mechanisms are involved in this pathophysiological process. Recent data demonstrated that remote, noninfarct-related region of the myocardium is also implicated. There is no data about the assessment of coronary endothelial function or myocardial fibrosis in the remote zone in patients with STEMI . The correlation between these parameters and left ventricular remodeling is not known.

ELIGIBILITY:
Inclusion Criteria:

* First ST Elevation Myocardial Infarction
* Primary Percutaneous Coronary Intervention (TIMI 3)
* Single vessel coronary artery disease
* Age over 18 years
* Informed Consent dated and signed
* Written and spoken French
* Beneficiary of social security insurance

Exclusion Criteria:

* No Primary Percutaneous Coronary Intervention
* TIMI 0-2 after Primary Percutaneous Coronary Intervention
* Significant two or three-vessel coronary artery disease (> 70% stenosis in at least one of the other two coronary arteries)
* Past history of myocardial infarction before STEMI
* Mechanical complication (ischaemic mitral regurgitation, interventricular septal defect, cardiac tamponade) or clinical signs of heart failure
* Pregnant and / or lactating
* Age under 18 years or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2022-08 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Measurement of coronary endothelial function | 3 months
  3 months following an acute coronary syndrome STEMI an ST segment (segments in myocardial infarcted area and "remote" ) .
Measurement of fibrosis | 3 months
  3 months following an acute coronary syndrome STEMI an ST segment (segments in myocardial infarcted area and "remote" ) .

SECONDARY OUTCOMES:
Correlating biomarkers with local and global parameters of coronary endothelial function , inflammation and myocardial fibrosis with early echocardiographic parameters of left ventricular remodeling and cardiac magnetic resonance imaging | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Farzin GF BEYGUI, PhD, Study Chair — CHU CAEN; Alain MA Manrique, PhD, Study Chair — CHU CAEN
Locations (1):
- CHu de Caen, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No